CLINICAL TRIAL: NCT06121141
Title: Comparison of Two Different Concentrations of Local Anesthetic in Patient Reported Pain in Oculoplastic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy Ekhlassi (Other)
Responsible Party: Sponsor-Investigator, Timothy Ekhlassi, Primary Investigator, Ekhlassi, Timothy, MD
Organization: Ekhlassi, Timothy, MD (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Thesis001
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Dermatochalasis; Dermatochalasis of Eyelid; Dermatochalasis of Both Upper Eyelids; Dermatochalasis of Both Eyes; Dermatochalasis of Right Upper Eyelid; Dermatochalasis of Left Upper Eyelid; Pain
Keywords: Dermatochalasis; Oculoplastic surgery; Eyelid surgery; Blepharoplasty; Upper blepharoplasty; Upper eyelid blepharoplasty
MeSH Terms: conditions — Cutis Laxa; Pain | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Full-strength lidocaine with epinephrine
  Interventions: Drug: Full strength lidocaine with epinephrine
- Experimental (Experimental): Dilute lidocaine with epinephrine
  Interventions: Drug: Dilute lidocaine with epinephrine

INTERVENTIONS:
Drug: Full strength lidocaine with epinephrine — 2% lidocaine with epinephrine 1:100,000
  Arms: Control
Drug: Dilute lidocaine with epinephrine — 2% lidocaine with epinephrine 1:100,000 diluted with normal saline (09.% NaCl) in a 1:4 ratio
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to compare pain scores in people undergoing upper eyelid surgery. The main questions it aims to answer are:

* Is one concentration of local anesthetic (also called numbing or freezing injection) less painful when it is injected?
* Does one concentration of local anesthetic provide better pain control during surgery? Participants will have two different concentrations of local anesthetic injected into the upper eyelid skin prior to surgery, and will be asked to rate the pain they have during the injection. At the end of surgery, they will be asked to rate the pain they have during surgery.

Researchers will compare the pain scores to see if one of the concentrations is less painful during the injection and to see if one of the concentrations provides better pain control during surgery.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate the level of pain experienced during injection of dilute local anesthetic when compared to non-dilute local anesthetic for oculoplastic surgery. It will also evaluate the level of pain experienced during surgery when comparing dilute local anesthetic to non-dilute local anesthetic for oculoplastic surgery.

Study design:

Randomized, double-blind study of 30 patients undergoing elective bilateral upper eyelid blepharoplasty, for a total of 60 eyes having surgery. For each patient, one side will be injected using the control medication consisting of non-dilute 2% lidocaine with epinephrine 1:100,000, and the other side will be injected using the treatment medication consisting of 2% lidocaine with epinephrine 1:100,000 diluted with normal saline (09.% NaCl) in a 1:4 ratio with normal saline (1 cc of anesthetic to 4 cc of normal saline). The distribution of which eyelid (right versus left) receives each arm will be randomized and hidden from both the researcher and the patient. Identical syringes and hypodermic needles will be used for the treatment and control arms. Each patient will then be asked to rate the pain experienced during local anesthetic injection for each side using a 100 mm visual analog scale (VAS). At the end of surgery, each patient will be asked to rate the level of pain experienced during the surgery on each side using a blank version of the same scale. Patients will be followed up for their regular post-operative appointment 7-21 days after surgery.

Data (VAS pain scores) will be collected on paper from each patient and entered into an Excel format spreadsheet. The need for additional local anesthetic, as well as the rate of anesthetic infiltration, will also be recorded in this Excel file. All data will be deidentified by assigning each participant an alphanumeric code.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older undergoing primary bilateral upper eyelid blepharoplasty
* Consent and compliance with all aspects of the study protocol

Exclusion Criteria:

* Patients undergoing two different types of surgery on either side (example, blepharoplasty on one side and ptosis repair on the other)
* Patients under 18 years old
* Patient scheduled for upper eyelid blepharoplasty who has had previous upper eyelid ptosis repair or upper eyelid blepharoplasty
* Patient undergoing unilateral surgery
* Active local or systemic malignancy
* Concurrent inflammatory lesion of the upper eyelids
* Participant is pregnant or plans to become pregnant during the treatment period
* Participant is involved in a WorkSafe (worker's compensation), personal injury suit, or other legal matter related to their health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Pain during injection | Immediately after injection
  Each patient will be asked to rate the pain experienced during local anesthetic injection for each side using a 100 mm visual analog scale (VAS)

SECONDARY OUTCOMES:
Pain during surgery | Immediately after surgery
  Each patient will be asked to rate the pain experienced during surgery for each side using a 100 mm visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ekhlassi, MD, Principal Investigator — Fraser Valley Cataract and Laser
Locations (1):
- Fraser Valley Cataract and Laser, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No